CLINICAL TRIAL: NCT05757154
Title: Coffee for Optimal Metabolite Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Paulig Group (Unknown)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ChalmersUA
Record Dates: First submitted 2023-02-18; First posted 2023-03-07 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Coffee A (Experimental): Coffee type A. All intervention arms are coffee. Three different types of coffee is tested. Differences in type of bean, degree of roasting and preparation method.
  Interventions: Other: Diet
- Coffee B (Experimental): Coffee type B. All intervention arms are coffee. Three different types of coffee is tested. Differences in type of bean, degree of roasting and preparation method.
  Interventions: Other: Diet
- Coffee C (Experimental): Coffe type C. All intervention arms are coffee. Three different types of coffee is tested. Differences in type of bean, degree of roasting and preparation method.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — All intervention arms are coffee. Three different types of coffee is tested. Differences in type of bean, degree of roasting and preparation method.

SUMMARY:
The aim of this project is to evaluate metabolite profile after consumption of three types of coffee differing in type of bean, degree of roasting and preparation method. Metabolite profiles will be evaluated after a) a single dose b) 3-day consumption. The study will be carried out as a three-way cross-over design with three different types of coffee. Wash-out periods where participants consume their habitual diet are implemented between all intervention periods. The first day of intervention (single dose) includes postprandial measurements during 13 hours.

ELIGIBILITY:
Inclusion Criteria:

* Females and males
* 18 to 80 years of age
* Body mass index (BMI) 18.5-30.0 kg/m2
* Fasting glucose ≤ 6.1 mmol/l
* Low density lipoprotein (LDL) cholesterol ≤ 5.30 mmol/l
* Triglycerides ≤ 2.60 mmol/l
* Signed informed consent

Exclusion Criteria:

* Food allergies or intolerances preventing consumption of any products included in the study.
* Unable to sufficiently understand written and spoken Swedish to provide written consent and understand information and instructions from the study personnel.
* Pregnant, lactating or planning a pregnancy during the study period.
* Antibiotic use for the last 3 months.
* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study.
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Chron's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* Previous major gastrointestinal surgery
* Have type I diabetes
* Thyroid disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 24 hours
  Difference in the plasma concentrations between the different types of coffee comparing before (baseline) and after single dose intervention.
Plasma concentration-time profile over 24 hours (AUC) of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 24 hours
  Difference in plasma AUC between the different types of coffee for each biomarker candidate.
Urine concentrations of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 24 hours
  Difference in the urine concentrations between the different types of coffee comparing before (baseline) and after single dose intervention.
Plasma kinetic profiles of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 24 hours
  Cmax will be estimated.
Plasma kinetic profiles of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 24 hours
  Tmax will be estimated.

SECONDARY OUTCOMES:
Plasma concentrations of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 4 days
  Difference in the plasma concentrations between the different types of coffee comparing before (baseline) and after single dose and three days intervention.
Urine concentrations of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 4 days
  Difference in the urine concentrations between the different types of coffee comparing before (baseline) and after single dose and three days intervention.
Plasma metabolites | 4 days
  Untargeted metabolomics will be performed using established methods for plasma. Analyzed exploratorily using untargeted metabolomics to find potential biomarker panels that reflect coffee consumption. Baseline compared with after intervention products.
Urine metabolites | 24 hours
  Untargeted metabolomics will be performed using established methods for urine. Analyzed exploratorily using untargeted metabolomics to find potential biomarker panels that reflect coffee consumption. Baseline compared with after intervention products.
Gut microbiome | 4 days
  Fecal samples will analyzed for composition of the gut microbiome, baseline compared with after 4 days of intervention products.
Blood concentrations of key metabolites derived from chlorogenic acid, caffeine, trigonelline and diterpenes. | 13 hours
  Evaluate new simple sampling techniques using dried blood spots.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Dr, Principal Investigator — Chalmers University of Technology
Locations (1):
- University of Gothenburg, Department of Food and Nutrition and Sport Science, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No